CLINICAL TRIAL: NCT04546386
Title: Retinal Vascular Changes After Endoscopic Endonasal Pituitary Surgery During One Year's Follow up, by Optical Coherence Tomography Angiography
Brief Title: Long-term Follow up for Retinal Vascular Changes After Endoscopic Endonasal Pituitary Surgery.
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Principal Investigator, Federico II University
Other Study IDs: 1003/19
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Pituitary Adenoma
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic endonasal pituitary surgery — Surgical treatment consisted of an endoscopic endonasal approach using a rigid 0-degree endoscope, 18 cm in length and 4 mm in diameter

SUMMARY:
This study investigates the retinal vascular features, using optical coherence tomography angiography, in patients during one year's follow up after the endoscopic endonasal surgery to remove an intra-suprasellar pituitary adenoma compressing the optic nerve.

DETAILED DESCRIPTION:
The role of the optical coherence tomography angiography to detect the changes in retinal vascular networks in patients after 48 hours and 1 year from the endoscopic endonasal surgery to remove an intra-suprasellar pituitary adenoma compressing the optic nerve.

The optical coherence tomography angiography allows a detailed and quantitative analysis of the retinal vascular networks and to follow their changes over time.

ELIGIBILITY:
Inclusion Criteria:

* age older than 45 years
* diagnosis of pituitary adenoma
* treatment-naive with endoscopic endonasal pituitary surgery
* absence of other neurological disease
* absence of vitreoretinal and vascular retinal diseases

Exclusion Criteria:

* age younger than 45 years
* No diagnosis of pituitary adenoma
* previous treatment with endoscopic endonasal pituitary surgery
* presence of neurological disease
* presence of vitreretinal and vascular retinal diseases

Ages: 45 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The partecipants were older than 45 years and they underwent long term follow up after endoscopic endonasal pituitary surgery to remove pituitary adenoma.
  They did not present other neurological and ophthalmological diseases
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Study of vessel density of the retinal vascular network in patients underwent endoscopic endonasal pituitary surgery, by optical coherence tomography angiography, during long-term follow up. | one year
  To evaluate the changes in vessel density of the retinal vascular network 48 hours and 1 year after endoscopic endonasal pituitary surgery for the removal of an intra-suprasellar pituitary adenoma compressing the optic nerve, using optical coherence tomography angiography. The parameter analyzed by optical coherence tomography angiography was the vessel density of the retinal vascular network.

CONTACTS AND LOCATIONS:
Overall Officials: Gilda Cennamo, Principal Investigator — Federico II University
Locations (1):
- University of Naples "Federico II", Naples, Italy